CLINICAL TRIAL: NCT02978703
Title: Non Interventional, Observational, Multi-center Study to Evaluate the Efficacy and Safety of Fluticasone/Salmeterol (Rolenium / Elpenhaler Administration in Greek COPD Pattients
Brief Title: EvAluation of Clinical Effectiveness Of RoLenium Administered With Elpenhaler in Chronic Obstructive Pulmonary Disease (COPD) patientS in Daily Clinical Practice, in Greece
Acronym: AEOLOS
Status: Completed | Type: Observational
Sponsor: Elpen Pharmaceutical Co. Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 2016-HAL-EL-67
Record Dates: First submitted 2016-11-16; First posted 2016-12-01 (Estimated); Last update posted 2019-05-13 (Actual); Status verified 2018-01

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: COPD Pharmacologic Substance — COPD patients treated by Fluticasone / Salmetrol via Elpenhaler device

SUMMARY:
Observational study for the evaluation of clinical effectiveness in daily clinical practice of inhaled combination of propionic Fluticasone and Salmeterol in doses (500+50)mcg - Rolenium- administered with Elpenhaler device in approximately 2000 COPD (Chronic Obstructive Pulmonary Disease) patients with a FEV1 <50% predicted normal (pre-bronchodilator), a history of repeated exacerbations and who have significant symptoms despite regular bronchodilator therapy in Greece.

DETAILED DESCRIPTION:
The scientific Objectives are to study in the Greek population the real-life patient characteristics of patients selected for treatment with the inhaled combination of propionic Fluticasone and Salmeterol (500+50)mcg - Rolenium- administered with Elpenhaler device and the performance of this inhaled combination in terms of effectiveness and safety in approximately 2500 COPD (Chronic Obstructive Pulmonary Disease) patients with a FEV1 <50% predicted normal (pre-bronchodilator), a history of repeated exacerbations and who have significant symptoms despite regular bronchodilator therapy treated in Hospital and outpatient specialist ward settings, in the daily clinical practice

The primary endpoints for the study are:

• Change in FEV1, FVC, FEV1/FVC from baseline to 12 months (±2 weeks) from starting taking Rolenium®.

The Secondary endpoints for the study are:

* Change in lung function parameters from baseline to month 6 (±2 weeks) from start of Rolenium® treatment
* Incidence and frequency of exacerbations
* Hospitalizations due to COPD exacerbation
* Change in MRC Dyspnea index.
* Patient's satisfaction with the use of Elpenhaler device assessed with FSI 10 Questionnaire after 6 months and after 12 months (±2 weeks).
* Concomitant administration of inhaled bronchodilators
* ADRs during the treatment period (only via the post-marketing procedure). Methodology The study will be a purely observational, prospective study, collecting data on patient treated with the inhaled combination of propionic Fluticasone and Salmeterol (500+50) mcg,- administered with Elpenhaler device in Greece without any interference with the treatment practices of the physicians involved in the data collection. Thus patients will only be considered for inclusion after the decision has been taken to treat them with inhaled combination of propionic Fluticasone and Salmeterol (500+50) mcg administered with Elpenhaler device and no visits, diagnostic procedures or monitoring will take place which would not happen had the patient not been included in the study. This means that only data generated in usual daily clinical practice will be collected in the study, so that no extra examinations or study visits will take place due to the study. The study will not be comparative; only inhaled combination of propionic Fluticasone and Salmeterol (500+50)mcg,- administered with Elpenhaler device will be included. Consecutive patients who are to start the inhaled combination of propionic Fluticasone and Salmeterol (500+50) mcg,- administered with Elpenhaler device treatment shall be informed about the study and asked for consent. Following usual practice the patients will be followed after 6 months and after 12 months (±2 weeks) of the inhaled treatment.

The patients' selection criteria will be according to SmPC.

ELIGIBILITY:
Inclusion Criteria:

* patients selected for treatment with the inhaled combination of propionic Fluticasone and Salmeterol (500+50)mcg - Rolenium- administered with Elpenhaler device
* FEV1 <50% predicted normal (pre-bronchodilator),
* a history of repeated exacerbations who have significant symptoms despite regular bronchodilator therapy treated in Hospital outpatient specialist ward settings, in the daily clinical practice
* have signed informed consent
* be compliant with study procedures

Exclusion Criteria:

* - patients not selected for treatment with the inhaled combination of propionic
* FEV1 >50% predicted normal (pre-bronchodilator),
* no history of repeated exacerbations
* not signed informed consent
* will not be compliant with study procedures

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: COPD patients will be recruited in the study. The patients will be diagnosed with COPD with a FEV1 <50% predicted normal (pre-bronchodilator) in need of symptomatic treatment and a history of repeated exacerbations, who have significant symptoms despite regular bronchodilator therapy.
  The study will be conducted in about 100 sites in Greece. 5 study sites will be Hospitals and 75 study sites will be pulmonologists in private practice.
  The investigators will be Pulmonologists.
  Patients that are to start treatment with the inhaled combination of propionic Fluticazone and Salmeterol in doses (250+50)mcg, (500+50)mcg are eligible for inclusion in the study. In accordance with the approved labelling these patients should:
Sampling Method: Non-Probability Sample
Enrollment: 1730 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Efficacy assessed by Spirometry | 12 months
  Spirometry: Change in FEV1
Efficacy assessed by MRC dyspnea questionnaire | 12 months
  MRC Dyspnea questionnaire

SECONDARY OUTCOMES:
Safety assessed by number of exacerbations | 0,6,12 months
  Incidence of exacerbations
Patient Satisfaction assessed by FSI-10 questionnaire | 12 months
  FSI-10 questionnaire score per patient per study visit

CONTACTS AND LOCATIONS:
Overall Officials: Nikolaos Tzanakis, MD, Study Chair — University of Herakleion, Crete
Locations (2):
- Greece (2):
  - University Hospital of Crete, Heraklion, Crete
  - University Hospital of Herakleion, Heraklion

IPD SHARING:
Plan to Share IPD: No